CLINICAL TRIAL: NCT01806545
Title: A Phase 2, Single-blind, Randomized, Controlled, Multi-center Study to Evaluate the Efficacy and Safety of SRM003 (Vascugel®) in Improving the Rate of Arteriovenous Fistula Maturation and Use in Subjects Undergoing Surgery for Creation of an Arteriovenous Fistula for Hemodialysis Access
Brief Title: An Efficacy and Safety Study of SRM003 in the Treatment of Subjects Undergoing Creation of an Arteriovenous Fistula to Facilitate Hemodialysis Access
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AVF01-SRM003
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Arteriovenous Fistula
Keywords: Arteriovenous Fistula Surgery; Vascular Injury; Hemodialysis Access
MeSH Terms: conditions — Arteriovenous Fistula; Vascular System Injuries | interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SRM003 (Active Comparator): One time implant (2 SRM003 pieces) on surgery day. Post-surgery, up to 26 weeks follow-up for assessment of efficacy/safety.
  Interventions: Biological: SRM003
- Participating Site's standard practice (Other): Subjects will receive sites' standard practice treatment during the surgical procedure.
  Interventions: Other: Participating Site's standard practice

INTERVENTIONS:
Biological: SRM003 — One time implant (2 SRM003 pieces) on surgery day.
  Other Names: Allogeneic human aortic endothelial cells cultured in a gelatin matrix (Gelfoam®).
  Arms: SRM003
Other: Participating Site's standard practice — Subjects will receive sites' standard practice treatment during the surgical procedure.
  Arms: Participating Site's standard practice

SUMMARY:
A study to evaluate the efficacy of SRM003 treatment versus participating sites' standard practice treatment in improving the rate of AVF maturation and use in subjects with end-stage renal disease undergoing surgery for creation of an AVF to facilitate hemodialysis access.

It is hypothesized that when placed outside the blood vessel, the seeded SRM003 gelatin matrix containing endothelial cells can provide a continuous supply of multiple growth regulatory compounds to the underlying cells within the blood vessel, while being protected from the effects of blood flow in the vessel(s) or complications resulting from being in direct contact with the point of injury.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 years of age or older at the time of signing and dating informed consent (no upper age limit), can be male or female.
2. Subject who is of child bearing potential must agree to use adequate contraception for 6 months after randomization.
3. Subject must be currently undergoing hemodialysis or anticipating the start of hemodialysis and must require a new permanent, suitable access for the AVF creation in the upper extremity.
4. Subject must have a life expectancy of at least 26 weeks after randomization.
5. Subject must be able to understand and be willing to complete all study requirements.

Exclusion Criteria:

1. Subject is currently on an active organ transplant list from a deceased donor or is undergoing assessment and expects to be placed on the active organ or bone marrow transplant list within the next 26 weeks from surgery, or expects to receive a living donor organ or bone marrow within the next 26 weeks and is unwilling to change transplant list status to "hold" for 3 months after randomization.
2. Subject has had more than 1 access placement surgery (defined as a new access, not a revision) in the target limb.
3. Subject has medical conditions and diseases that may cause non-compliance with the protocol
4. Subject has a known allergy to bovine/porcine products or collagen/gelatin products.
5. Subject has a history of intravenous drug use within 6 months prior to screening
6. Subject is morbidly obese, defined as having a body mass index >40.
7. Pregnant or nursing woman, or plans to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-03-26 (Actual); Primary Completion 2014-10-27 (Actual); Study Completion 2014-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (47):
- United States (47):
  - Akdhc Medical Research Services, Phoenix, Arizona
  - Tucson Vascular Consultants, Tucson, Arizona
  - Ladenheim Dialysis Access Center, Fresno, California
  - California Institute of Renal Research, La Mesa, California
  - VA Long Beach Health Care System Pharmacy, Long Beach, California
  - The Regents University of California Los Angeles, Los Angeles, California
  - California Institute of Renal Research, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Tampa General Hospital, Tampa, Florida
  - Georgia Regents University, Augusta, Georgia
  - Illinois Kidney Disease & Hypertension Center, Peoria, Illinois
  - University of Louisville, Louisville, Kentucky
  - Ochsner Baptist Medical Center, Clinical Trials Unit, New Orleans, Louisiana
  - Louisiana State University Health Science Center Shreveport, Shreveport, Louisiana
  - Baystate Medical Center Pharmacy, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Renaissance Renal Research Institute, LLC, Detroit, Michigan
  - McLaren Northern Michigan Hospital-NISUS Research, Petoskey, Michigan
  - Providence Hospital, Research Dept., Southfield, Michigan
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Sierra Nevada Nephrology Consultants, Reno, Nevada
  - United Health Services, Johnson City, New York
  - Mount Sinai School of Medicine Lab, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Metrolina Nephrology Associates, PA, Charlotte, North Carolina
  - ECU Department of Nephrology and Hypertension, Greenville, North Carolina
  - Sanford Research/USD-Fargo, Fargo, North Dakota
  - University of Cincinnati Physicians Company, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Kaiser Permanente Northwest, Milwaukie, Oregon
  - Northwest Renal Clinic, Inc., Portland, Oregon
  - Penn Medicine, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Delaware Valley Nephrology and Hypertension Associates, PC, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - SC Nephrology & Hypertension Center, Inc., Orangeburg, South Carolina
  - Erlanger Hospital Pharmacy, Chattanooga, Tennessee
  - Nephrology Associates, P.C., Nashville, Tennessee
  - Baylor College of Medicine ICTR, Houston, Texas
  - Fletcher Allen Health Care Renal Service, Burlington, Vermont
  - Sentara Vascular Specialists, Norfolk, Virginia
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - University of Wisconsin, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Participating Site's Standard Practice: Participants received the site's standard practice treatment during the surgical procedure. Post-surgery, each participant was to undergo 26 weeks of follow-up for assessment of efficacy and safety.
- SRM003: Participants received a one-time implant of 2 SRM003 pieces on surgery day after the completion of the arteriovenous fistula (AVF) creation. One sponge was wrapped around the venous anastomosis site and the other was placed longitudinally on the vein segment, immediately distal to the venous anastomosis. Subjects were not permitted to undergo additional applications with SRM003 sponges after the initial application. Post-surgery, each participant was to undergo 26 weeks of follow-up for assessment of efficacy and safety.
Period: Overall Study
Arm/Group | Participating Site's Standard Practice | SRM003
Started | 29 | 35
Completed | 23 | 30
Not Completed | 6 | 5
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: The Intent -to-Treat (ITT) population, defined as all randomly assigned participants regardless of receiving treatments or having post-baseline outcome data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participating Site's Standard Practice | SRM003 | Total
Number analyzed (Participants) | 29 | 35 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (13.5) | 61.1 (10.8) | 63.0 (12.2)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 12 | 23 | 35
  ≥65 years | 17 | 12 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Arteriovenous Fistula (AVF) Maturation by Week 12 Visit Based on Hemodialysis or Color-flow Doppler Ultrasound (CDUS) And Vascular Access Examination
Description: Maturation based on CDUS was assessed in a continuous fashion and was defined by the following criteria: presence of bruit throughout systole and diastole at least 8 centimeters (cm) proximal to the venous anastomosis, blood flow through the outflow vein of at least 500 milliliters (ml) per minute, and a lumen diameter of the outflow vein at least 4 mm. Maturation was determined by CDUS and vascular access examination or by first use of the AVF for hemodialysis based on investigator-reported use. Participants who discontinued prior to the Week 12 visit without assessment of maturity were considered treatment failures.
Time Frame: 12 weeks after surgery
Population: The Intent- to-Treat (ITT) population, defined as all randomly assigned participants regardless of receiving treatments or having post-baseline outcome data.
Measure: Number; unit: percentage of participants
Arm/Group | Participating Site's Standard Practice | SRM003
Number analyzed (Participants) | 29 | 35
percentage of participants | 96.6 | 85.7
Statistical Analysis 1: Comparison: Participating Site's Standard Practice vs SRM003; Test type: Superiority or Other; p = 0.1197, Cochran-Mantel-Haenszel — P-value was based on Cochran-Mantel-Haenszel test stratified by diabetic status at surgery comparing the 2 treatment groups; Proportion treatment difference = -0.11, 95% CI 2-sided [-0.242 to 0.025]

2. Secondary Outcome: Percentage of Participants With AVF Maturation by Week 26 Visit Based on Hemodialysis or CDUS And Vascular Access Examination
Description: Maturation based on CDUS was assessed in a continuous fashion and was defined by the following criteria: presence of bruit throughout systole and diastole at least 8 centimeters (cm) proximal to the venous anastomosis, blood flow through the outflow vein of at least 500 milliliters (ml) per minute, and a lumen diameter of the outflow vein at least 4 mm. Maturation was determined by CDUS and vascular access examination or by first use of the AVF for hemodialysis based on investigator-reported use. Participants who discontinued prior to the Week 26 visit without assessment of maturity were considered treatment failures.
Time Frame: 26 weeks after surgery
Population: The ITT population, defined as all randomly assigned participants regardless of receiving treatments or having post-baseline outcome data.
Measure: Number; unit: percentage of participants
Arm/Group | Participating Site's Standard Practice | SRM003
Number analyzed (Participants) | 29 | 35
percentage of participants | 96.6 | 88.6
Statistical Analysis 1: Comparison: Participating Site's Standard Practice vs SRM003; Test type: Superiority or Other; p = 0.1962, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Proportion treatment difference = -0.08, 95% CI 2-sided [-0.204 to 0.045]

3. Secondary Outcome: Time to AVF Maturation Based on Hemodialysis or CDUS and Vascular Access Examination
Description: Time to AVF maturation was defined as the duration of time (in days) from the date of randomization (AVF creation) to the date of maturation, where the date of maturation corresponds to the earlier of either the date of the first use of the study AVF for hemodialysis as determined by the investigator following discussion with the participant, or the date the AVF meets all of the following 3 criteria as determined through CDUS and vascular access examination: presence of bruit throughout systole and diastole at least 8 centimeters proximal to the venous anastomosis, blood flow through the outflow vein of at least 500 milliliters (ml) per minute, and a lumen diameter of the outflow vein at least 4 mm. Participants who died, underwent a kidney transplant, or were either lost to follow-up or did not mature during the study follow-up were censored at the time of death, time of transplant, or time of last visit, respectively.
Time Frame: Up to 26 weeks after surgery
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Participating Site's Standard Practice | SRM003
Number analyzed (Participants) | 29 | 35
days | 9 [8 to 28] | 10 [8 to 59]
Statistical Analysis 1: Comparison: Participating Site's Standard Practice vs SRM003; Test type: Superiority or Other; p = 0.090, Log Rank — P-value based on log-rank test stratified by diabetic status at surgery comparing the 2 treatment groups

4. Secondary Outcome: Percentage of Participants With Loss of Unassisted Primary Patency
Description: The time to loss of unassisted primary patency (intervention--free access survival) was defined as the duration of time in days from the date of randomization (AVF creation) until the first date of (a) any intervention designed to establish, maintain, or restore patency; (b) occlusion (commonly due to thrombosis); or (c) access abandonment.
Time Frame: Up to 26 weeks after surgery
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Participating Site's Standard Practice | SRM003
Number analyzed (Participants) | 29 | 35
percentage of participants | 20.7 | 37.1
Statistical Analysis 1: Comparison: Participating Site's Standard Practice vs SRM003; Analysis of time to loss of patency; Test type: Superiority or Other; p = 0.193, Log Rank; P-value based on log-rank test stratified by diabetic status at surgery comparing the 2 treatment groups

5. Secondary Outcome: Percentage of Participants With Loss of Assisted Primary Patency
Description: The time to loss of assisted primary patency (thrombosis--free access survival) was defined as the duration of time in days from the date of randomization (AVF creation) until the first date of (a) occlusion (commonly due to thrombosis) or (b) access abandonment.
Time Frame: Up to 26 weeks after surgery
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Participating Site's Standard Practice | SRM003
Number analyzed (Participants) | 29 | 35
percentage of participants | 6.9 | 17.1
Statistical Analysis 1: Comparison: Participating Site's Standard Practice vs SRM003; Analysis of time to loss of patency; Test type: Superiority or Other; p = 0.231, Log Rank — P-value based on log-rank test stratified by diabetic status at surgery comparing the 2 treatment groups

6. Secondary Outcome: Percentage of Participants With Loss of Secondary Patency
Description: The time to loss of secondary patency (access survival until abandonment) was defined as the duration of time in days from the date of randomization (AVF creation) until the date of access abandonment.
Time Frame: Up to 26 weeks after surgery
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Participating Site's Standard Practice | SRM003
Number analyzed (Participants) | 29 | 35
percentage of participants | 3.4 | 14.3
Statistical Analysis 1: Comparison: Participating Site's Standard Practice vs SRM003; Analysis of time to loss of patency; Test type: Superiority or Other; p = 0.158, Log Rank — P-value based on log-rank test stratified by diabetic status at surgery comparing the 2 treatment groups

7. Secondary Outcome: Change From Week 1 in Average Vascular Access Lumen Diameter Using CDUS
Description: B-mode lumen diameter measurements were obtained in the outflow vein as 3 separate images for each location: at 1, 3, and 5 centimeter into the vein and from the toe of the venous anastomosis. The average of lumen diameter measurements obtained at 1, 3, and 5 cm from the anastomosis was used for this endpoint.
Time Frame: 1, 12, and 26 weeks after surgery
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Participating Site's Standard Practice | SRM003
Number analyzed (Participants) | 29 | 35
millimeters
  Week 12, n=21, 28 | 1.897 (1.2587) | 1.253 (1.9908)
  Week 26, n=20, 25 | 2.489 (1.4525) | 2.416 (2.3941)
Statistical Analysis 1: Comparison: Participating Site's Standard Practice vs SRM003; Treatment difference at week 12; Test type: Superiority or Other; Mean treatment difference = -0.895, 95% CI 2-sided [-2.213 to 0.423]
Statistical Analysis 2: Comparison: Participating Site's Standard Practice vs SRM003; Treatment difference at week 26; Test type: Superiority or Other; Mean treatment difference = -0.232, 95% CI 2-sided [-1.791 to 1.327]

8. Secondary Outcome: Percentage of Participants With Clinical Success Based on First Use of The Study AVF For Hemodialysis
Description: Clinical success was defined as the ability to undergo hemodialysis using the AVF. The date of clinical success corresponded to the date of the first use of the study AVF for hemodialysis as determined by the investigator, following discussion with the subject. Clinical success was assessed in a continuous fashion and, once achieved, the AVF was considered a clinical success at that and all subsequent time points. The date of clinical success based on the first use of the AVF for hemodialysis was compared with the dates of each study visit (Week 12 and Week 26); for study visits occurring prior to the date of clinical success based on the first use of the AVF for hemodialysis, the subject was counted as a nonsuccess and for study visits occurring on or after the date of maturation based on the first use of the AVF for hemodialysis, the subject was counted as a success.
Time Frame: 12 and 26 weeks after surgery
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Participating Site's Standard Practice | SRM003
Number analyzed (Participants) | 29 | 35
percentage of participants
  Week 12 | 37.9 | 34.3
  Week 26 | 55.2 | 62.9
Statistical Analysis 1: Comparison: Participating Site's Standard Practice vs SRM003; Analysis of week 12; Test type: Superiority or Other; Proportion treatment difference = -0.04, 95% CI 2-sided [-0.273 to 0.200]
Statistical Analysis 2: Comparison: Participating Site's Standard Practice vs SRM003; Analysis of week 26; Test type: Superiority or Other; Proportion treatment difference = 0.08, 95% CI 2-sided [-0.165 to 0.318]

9. Secondary Outcome: Number of Interventions to Establish, Maintain, or Restore Patency
Description: The total number of interventions to establish, maintain, or restore patency was recorded for each participant.
Time Frame: 12 and 26 weeks after surgery
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: interventions
Arm/Group | Participating Site's Standard Practice | SRM003
Number analyzed (Participants) | 29 | 35
interventions
  Week 12 | 0.1 (0.31) | 0.3 (0.61)
  Week 26 | 0.2 (0.49) | 0.8 (1.52)
Statistical Analysis 1: Comparison: Participating Site's Standard Practice vs SRM003; Analysis of week 12; Test type: Superiority or Other; Mean treatment difference = 0.154, 95% CI 2-sided [-0.096 to 0.404]
Statistical Analysis 2: Comparison: Participating Site's Standard Practice vs SRM003; Analysis of week 26; Test type: Superiority or Other; Mean treatment difference = 0.565, 95% CI 2-sided [-0.023 to 1.152]

ADVERSE EVENTS:
Description: Treatment emergent adverse events are presented for the safety population, defined as all randomly assigned participants who received either SRM003 treatment or participating sites' standard practice treatments.
Arm/Group | Participating Site's Standard Practice | SRM003
Serious Adverse Events (participants affected / at risk) | 16/29 | 13/35
Other Adverse Events (participants affected / at risk) | 17/29 | 25/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participating Site's Standard Practice (N=29) | SRM003 (N=35)
Acute myocardial infarction (Cardiac disorders) | 2 (3) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Non cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 1 (3)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 3 (3)
Steal syndrome (Vascular disorders) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participating Site's Standard Practice (N=29) | SRM003 (N=35)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 0 (0) | 3 (3)
Local swelling (General disorders) | 2 (2) | 3 (3)
Medical device complication (General disorders) | 0 (0) | 3 (5)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 5 (8) | 7 (12)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 4 (5) | 2 (3)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Renal failure chronic (Renal and urinary disorders) | 2 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually